CLINICAL TRIAL: NCT05692258
Title: Acupuncture as an Adjunctive Therapy for Covid-19 Omicron Randomised Controlled Trial in Patients With Moderate/Severe Pneumonia
Acronym: ZCFZZLXGBDFYHZ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, ZhangWei, The First Affiliated Hospital of Hunan University of Chinese Medicine, The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019SK4004-06
Record Dates: First submitted 2023-01-17; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Acupuncture; Covid-19 Omicron; Pulmonary Function
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled study. According to the design of stratified random grouping, the subjects is stratified according to the degree of disease (moderate, severe) and age stage (30-59 years, > 60 years), and then randomly assigned to the observation group and the control group within each stratum.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: On account of the particularity of acupuncture research, it is impossible to blind acupuncture operators. Blinded evaluation will be adopted in the trial, and the third party who does not know the grouping will evaluate the efficacy. Blind statistical analysis was used in the data summary stage, and the researchers, operators and statisticians were separated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture therapy + basic therapy (Experimental): Acupuncture treatment-Selected acupoints: Dazhui (GV14) , Feishu(BL13), Dingchuan(EX-B1), Tiantu(CV22), Danzhong(RN17), Quchi(LI11), Kongzui(LU6), Neiguan(PC6), Yinlingquan(SP9), Fenglong(ST40), Qihai(cv6). Once a day for 10 consecutive times.
  Western medicine treatment (basic treatment) : According to the Diagnosis and Treatment Plan for Novel Coronavirus Infection (Trial 10th Edition) issued by the General Office of the National Health Commission and the General Department of the National Administration of Traditional Chinese Medicine, patients are arranged to be quarantined in hospitals for treatment. Conventional Western medicine treatment includes supportive treatment, antiviral therapy, immunotherapy, anticoagulant therapy, antibiotic therapy, etc.
  Interventions: Other: Acupuncture
- sham acupuncture + basic therapy (Sham Comparator): sham acupuncture. Acupoint selection, body position, intervention time and course of treatment are the same as those in acupuncture treatment group. After acupoint disinfection, fixed pad is pasted on the acupoint, and 1.5 blunt needle will be used to Pierce directly through the sham instrument to fix pad to the skin surface without piercing the skin, and do not require Deqi. Western medicine treatment (basic treatment) is the same as the acupuncture group.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture is a kind of therapy used to treat diseases, in which a needle (usually a millimeter needle) is inserted into a patient's skin or tissue at a certain Angle to stimulate a specific part of the body (acupoint).
  Disposable sterile acupuncture filiform needle (0.30mm×25mm、0.30mm×40mm), Guizhou Andi Medical Equipment Co, LTD, Guizhou Food and Drug Supervision and Equipment Production Xu 20170011.
  Other Names: basic therapy

SUMMARY:
At present, China is facing the first wave of COVID-19 epidemic after the liberalization. The infection rate has exceeded 50% in most areas, and even exceeded 80% in some cities. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) belongs to the beta genus of coronavirus and enters cells mainly by binding angiotensin converting enzyme 2 (ACE-2) to the spike protein on the envelope. The Omicron strain is the main epidemic strain at present. The transmission ability of Omicron strain is stronger than Delta strain, but the pathogenicity is weakened. At present, the published articles on the adjuvant treatment of COVID-19 with acupuncture are mostly theoretical discussions or case reports, and randomized controlled trials on the observation of curative effect are rare. The purpose of this study is to clarify the effectiveness of the adjuvant treatment of COVID-19 with acupuncture. Providing high-level research evidence for them.

DETAILED DESCRIPTION:
This is a stratified randomized trial. Firstly, the subjects were stratified according to disease severity (moderate, severe) and age stage (30-59 years, > 60 years), and then the subjects were randomly assigned to the observation group and the control group within each stratum. The study center will screen cases strictly according to the diagnostic criteria, inclusion criteria and exclusion criteria. After confirmation of enrollment, random numbers will be obtained according to the application for random coding process until the total number of observation is completed. Blinded evaluation will be adopted in the trial, and the third party who does not know the grouping will evaluate the efficacy. Blind statistical analysis was used in the data summary stage, and the researchers, operators and statisticians were separated. In the observation group (acupuncture treatment + basic treatment), acupuncture will be applied at Dazhui (GV 14), Feishu (BL 13), Dingchuan (GV 14), Tiantu (GV 14), Danzhong (CV 17), Quchi (GV 20), Gongzhi (CV 4), Neiguan (PC 6), Yinlingquan (SP 9), Fenglong (ST 40), Qihai (CV 6). In the control group (sham acupuncture + basic treatment), sham acupuncture will be used. The acupoint selection is the same as the acupuncture treatment group, Before acupuncture, the fixed pad was pasted on the acupoints, 1.5-inch blunt needle will be used to Pierce the skin surface through the fixed pad of the sham appliance without puncturing the skin.

The mMRC and COVID-19 symptom assessment scale were used as the main evaluation indicators, and the Leicester cough questionnaire LCQ was used to record cough. VAS pain score visual analogue scale was used to evaluate the daily situation of sore throat, muscle soreness, and headache. Secondary outcomes included vital signs and oxygen saturation, chest CT score, and related blood biochemical indicators, including: Blood routine, coagulation routine, D-dimer, C-reactive protein, erythrocyte sedimentation rate, procalcitonin, cytokines (interleukin-6, interleukin-1, ferritin), myocardial enzymes, T lymphocyte subsets (CD4+, CD8+), liver function, renal function, blood gas analysis (severe patients), nucleic acid negative conversion rate, severe conversion rate, self-rating anxiety scale (SAS). Uniform training was provided to all study personnel. The training focused on the use of randomization system and case entry system, project implementation and standard operating procedures, so that each researcher could be familiar with the research process and specific implementation rules, so as to improve the intra-observer consistency and inter-observer consistency of researchers and ensure the reliability of clinical research conclusions. An independent efficacy evaluator was required. Efficacy raters and statistical analysts were blinded. Statistical analyses were performed by a third party, and statistical analysts were blinded during the trial. Statistical analysis will be calculated using SPSS22.0 statistical analysis software. P<0.05 (i.e., =0.05) was considered to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* (1) in accordance with the diagnostic criteria of western medicine. (2) moderate and severe clinical types; (3) patients over 30 years old. (4) Patients voluntarily participated in the study and signed the informed consent.

Exclusion Criteria:

- (1) critical COVID-19 patients; (2) Allergic constitution, allergic to traditional Chinese medicine components; (3) pregnant or lactating women; (4) complicated with severe cognitive and mental disorders that cannot be clearly expressed; (5) those participating in other clinical trials; (6) According to the investigator's judgment, there will be patients with complicated enrollment or poor compliance, which will affect the efficacy and safety evaluation.

(7) complicated with active pulmonary tuberculosis, malignant arrhythmia, acute myocardial infarction, acute stroke, etc.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-04-06 (Estimated); Study Completion 2023-04-06 (Estimated)

PRIMARY OUTCOMES:
Modified Medical Research Council Dyspnea Scale | Once a day
  On a scale of 0-4, the higher the score, the more severe the symptoms
Symptom Assessment Scale for novel coronavirus pneumonia | Evaluate once a day
  15 items: 7 main symptoms (0-3 points), 8 secondary symptoms (0-1 points), the higher the score, the more severe the symptoms
Leicester cough questionnaire | During the screening period and on the 10th day of treatment
  19 items, divided into physiological, pathological and social dimensions, each item scored 1-7 points. Dimension score = Total score of item questions in each dimension ➗ Number of questions (1-7).Total score = Sum of three dimensions scores (3-21)
Visual Analogue Scale/Scor | Evaluate once a day
  3 items: pharyngeal pain, muscle soreness, headache. Pain is divided into 10 points, 0 points means no pain, 10 points means severe pain, the middle part of the different degrees of pain. Have the patient draw a mark on the horizontal line according to how they feel, which indicates the level of pain. The higher the score, the worse the pain.

SECONDARY OUTCOMES:
Vital signs and oxygen saturation | Record twice daily
  Body temperature, pulse, respiration, blood pressure, oxygen saturation
Chest CT score | Screening period, the 10th day of treatment
  In 6 areas of the right lung upper field, right lung middle field, right lung lower field, left lung upper field, left lung middle field, left lung lower field, reticular change 1 point, ground glass 2 points, patchy blur 3 points, small patchy blur 4 points, cystic lung honeycomb 5 points, the total score is 30 points, the higher the score is, the more severe the lung lesions.
Related blood biochemical indicators | Screening period, treatment days 3, 7, and 10.
  Routine blood test, coagulation test, D-dimer, C-reactive protein, erythrocyte sedimentation rate, procalcitonin, cytokines (interleukin-6, interleukin-1, ferritin), myocardial enzymes, T lymphocyte subsets (CD4+, CD8+), liver function, renal function laboratory indicators, and blood gas analysis were also recorded in severe patients.
Negative conversion rate of nucleic acid | Screening period, treatment days 3, 7, and 10.
  The nucleic acid of 2019-ncov will be detected by fluorescence quantitative polymerase chain reaction, and the negative conversion rate of nucleic acid will be calculated
Conversion rate of severe disease | Tenth day of treatment
  According to the clinical classification of "Diagnosis and Treatment Protocol for Novel Coronavirus Infection (Trial 10th Edition)", the number of patients who turned from medium to severe or critical will be recorded. Calculate the conversion rate of severe disease (number of severe disease cases/total cases × 100%)
The total score of the self-rating anxiety Scale | Screening period, treatment days 3, 7, and 10
  20 items, each item 1-4 points, total score and standard score (total score ×1.25), the higher the score, the more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Doctor, Study Chair — +86 135 4863 9198
Locations (1):
- The First Affiliated Hospital of Hunan University of Chinese Medicine, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Our subject database is called Zintuikang Integrated Big Data Application Platform, and other researchers can access it through the website. The administrator set up the account, and other researchers can log in by changing the password after registration. Their account has the authority to access the data and enter the CRF form.

REFERENCES:
- [Result] Liu ST, Zhan C, Ma YJ, Guo CY, Chen W, Fang XM, Fang L. Effect of qigong exercise and acupressure rehabilitation program on pulmonary function and respiratory symptoms in patients hospitalized with severe COVID-19: a randomized controlled trial. Integr Med Res. 2021;10(Suppl):100796. doi: 10.1016/j.imr.2021.100796. Epub 2021 Oct 29. PMID 34733607
- See also: Chen Wen-tao, Fu Huai-li, ZHANG Chao-yuan, et al. Feasibility Analysis of Acupuncture and Moxibustion in the Prevention and Treatment of COVID-19 from an International Perspective. Clinical Journal of Acupuncture and Moxibustion, 2020, 36(9): 82-87. — http://kns.cnki.net.hnucm.opac.vip/KXReader/Detail?invoice=gze5UIE9Q3FuCnOu1YRN%2BiCwI2UI2UCZvAtrR0fHKxDfVyMfBw8Arl0qAA1f2cH2yhnOUracq8Ij7i5TLwzzsOikj7MqShZ2RZB6y3soW9qXFNFKHlqS88zPDo%2FhumNHMkTN35znxkjWlDt94nOZB4eAE3ZdrUqGxHOLFhYbkmg%3D&DBCODE=CJFD&FileName=ZJLC202009021&TABLEName=cjfdlast2020&nonce=2264F64B440C4602A8D2E12DB11E3E2B&uid=&TIMESTAMP=1673599446541
- See also: Gong Yabin, Shi Xin-jie, Zhang Yan, et al. Clinical application and practice ofacupuncture therapy in treatment of coronavirus disease 2019. Chinese Acupuncture and Moxibustion, 2021, 41(2): 142-144. — http://kns.cnki.net.hnucm.opac.vip/KXReader/Detail?invoice=hJnoZj%2BwVzUzyXuOanIy0k%2Frb8wPX27e1oMnetz6JwfjapXJKdSZcx8zsW3PPc8gfQf9g5%2B7TBwG%2FJV6cUACmxsi4xTTZDDBNAMp69vwAZ69inEeh3bfpM0biWZhD23TL%2BO9nQ0hBxBaNsNUc76iM29n569ygwJJEW74r2XdfOY%3D&DBCODE=CJFD&FileName=ZGZE202102009&TABLEName=cjfdlast2021&nonce=54B21AEDF168419FB99D068D6564ADA5&uid=&TIMESTAMP=1673599706418
- See also: Yin Xin, CAI Shubin, Chen Luming, et al. Seventeen cases with coronavirus disease 2019(COVID-19)treated with the combination of acupuncture and herbal medicine. Chinese Acupuncture and Moxibustion, 2021, 41(5): 498-500. — http://kns.cnki.net.hnucm.opac.vip/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFDLAST2021&filename=ZGZE202105007&uniplatform=NZKPT&v=ymNwlExQ0p8iVITbnlr7LmEbS-Z8sA-uPSCEYTABJHzI1r5snIrG3n8TflNU_-Bu
- See also: Diagnosis and Treatment Protocol for Novel Coronavirus infection (Trial version 10) — http://www.gov.cn/zhengce/zhengceku/2023-01/06/content_5735343.htm